CLINICAL TRIAL: NCT04267926
Title: MitoQ for Fatigue in Multiple Sclerosis: A Placebo Controlled Trial
Brief Title: MitoQ for Fatigue in Multiple Sclerosis (MS)
Acronym: MitoQ
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURB-022-19S; 4337 (Other Grant/Funding Number: CSR&D)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Multiple Sclerosis; Fatigue; Mitochondrial
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — mitoquinone; mitoquinol

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized trial
Who Masked: Participant, Investigator
Masking Description: The subject and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 20mg of MitoQ (Active Comparator): 20mg of oral mitoquinol
  Interventions: Drug: 20 mg MitoQ
- 40mg of MitoQ (Active Comparator): 40mg of Oral Mitoquinol
  Interventions: Drug: 40mg of MitoQ

INTERVENTIONS:
Drug: 20 mg MitoQ — a third of subject will receive 20mg of oral MitoQ
  Other Names: Oral Mitoquinol
  Arms: 20mg of MitoQ
Drug: Placebo — Subject will receive Placebo
  Arms: Placebo
Drug: 40mg of MitoQ — a third of subjects will receive 40mg of MitoQ
  Other Names: Oral Mitoquinol
  Arms: 40mg of MitoQ

SUMMARY:
The purpose of this study is to determine whether MS patients who receive Oral mitoquinone (MitoQ) have less fatigue than those receiving a placebo. A comparison between patient's fatigue scored at baseline and fatigue scored 12 weeks after drug initiation will assess if MitoQ has a significant change in fatigue.

DETAILED DESCRIPTION:
Recruitment of subjects on hold due to COVID-19 pandemic

MitoQ is a potent antioxidant dietary supplement with potentially significant immunomodulatory and anti-inflammatory properties. While the cause of MS related fatigue is uncertain, the investigators believe that mitochondria dysfunction and resultant neuronal energy depletion may be an important contributor to fatigue in MS.

This clinical trial will evaluate the potential beneficial effects of MitoQ on MS fatigue. It will also explore the effects of MitoQ on cognitive function, quality of life and mood. If enrolled in the study, patients will take two capsules of the study drug or placebo at the same time every day for twelve weeks. There will be 4 study visits where the participant will undergo medical and nervous system examinations, questionnaires, and blood draws. Because it is a placebo-controlled trial, participants will have a 33% chance of receiving either placebo (inactive), 20mg of MitoQ, or 40mg of MitoQ. This will be a blinded randomized study, meaning neither the participant nor the investigator will know who received the placebo or study drug.

ELIGIBILITY:
Inclusion Criteria:

* MS (any clinical subtype) as diagnosed by the 2017 McDonald criteria
* EDSS score of 2 to 8
* complaint of fatigue that has been persistent for at least two months
* Modified Fatigue Impact Scale (MFIS) score of 38 or greater

Exclusion Criteria:

* treatment with systemic glucocorticoids in the prior six weeks
* Beck Depression Inventory (BDI) >31 or BDI-FS>10 (severe depression)
* significant MS exacerbation in prior 30 days
* previous use of MitoQ or Coenzyme Q10 (CoQ10) within thirty days of screening appointment
* other significant health problem that might increase risk of patient experiencing Adverse Events (AEs), e.g.:

  * active coronary heart disease
  * liver disease
  * pulmonary disease
  * diabetes mellitus
* pregnancy or intending to become pregnant or breastfeeding
* unable to complete the self-report forms
* unable to give informed consent
* prisoners
* any condition which would make the patient in the opinion of the investigator unsuitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, MBBS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen at the Multiple Sclerosis at Portland VA Medical Center (PORVAMC)and Oregon Health & Science University (OHSU) were main sources of recruitment. PORVAMC and OHSU MS clinics neurologists' referrals, chart reviews of MS patients at PORVAMC and OHSU Electronic medical records using the Mychart tool were used for help with recruitment. We additionally reached to a wide network of interested referring physicians from Portland and its surrounding areas.
Pre-assignment Details: Out of 46 screened subjects, 45 were randomized. One subject was NOT randomized due to abnormal screening labs. Two subjects were excluded after randomization (one subject had abnormal screening labs, second subject received IV Iron infusion for anemia). Thus, data from 43 subjects is available for the statistical analysis.
Groups:
- Placebo: Capsule containing Placebo ingredient.
- 20 mg of MitoQ: This group received one pill of the placebo and the second pill containing 20 mg of oral Mitoquinol (active drug) by mouth. Study drug was given empty stomach as described in the protocol.
- 40mg of MitoQ: This group received two pills, each containing 20 mg of oral Mitoquinol (active drug) thus total dose of 40 mg Mitoquinol, by mouth. Study drug was given empty stomach as described in the protocol.
Period: Overall Study
Arm/Group | Placebo | 20 mg of MitoQ | 40mg of MitoQ
Started | 16 | 15 | 14
Completed | 15 | 15 | 13
Not Completed | 1 | 0 | 1
Not completed — abnormal labs. No longer eligible | 0 | 0 | 1
Not completed — Iron infusion for fatigue. No longer eligible for study. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 20mg of MitoQ | 40mg of MitoQ | Total
Number analyzed (Participants) | 16 | 15 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age, Continuous
  Years | 54.8 (8.46) | 55.7 (9.32) | 52.6 (12.06) | 54.42 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 34
  Male | 4 | 3 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 16 | 15 | 13 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Modified Fatigue Inventory Scale (MFIS)
Description: MFIS is a self - reported fatigue survey. Scale 0 - 84. Higher scores indicate a greater impact of fatigue.
Time Frame: Week 1, Week 7, Week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 20mg of MitoQ | 40mg of MitoQ
Number analyzed (Participants) | 16 | 15 | 14
units on a scale
  Week 1 | 46.5 (2.8) | 55.2 (2.8) | 54.3 (2.9)
  Week 7 | 45.1 (3.1) | 50.5 (2.9) | 49 (3.1)
  Week 13 | 39.7 (2.8) | 48.7 (2.8) | 47.8 (3)
Statistical Analysis 1: Comparison: Placebo vs 20mg of MitoQ vs 40mg of MitoQ; Test type: Other; p = 0.9489, Mixed Models Analysis; In our work there are several hypotheses for the group comparison for the change. Therefore multiple estimate values that are not suitable for the questions above

2. Secondary Outcome: Symbol Digit Modalities Test (SDMT)
Description: SDMT measures cognitive function. Scale 0-110. Higher scores reflect a better outcome.
Time Frame: Week 1, Week 7, Week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 20mg of MitoQ | 40mg of MitoQ
Number analyzed (Participants) | 16 | 15 | 14
units on a scale
  Week 1 | 31.3 (8.4) | 25.9 (8.1) | 33.3 (8.4)
  Week 7 | 33.2 (8.0) | 28.8 (8.0) | 36.1 (8.2)
  Week 13 | 32.6 (8.4) | 30.4 (8.1) | 35.6 (8.2)

3. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: EDSS measures neurological function. Scale 0-10
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Beck's Depression Inventory (BDI)
Description: BDI is a self-reported questionnaire measuring depression. Scale 0-21
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up (13 weeks)
Arm/Group | Placebo | 20mg of MitoQ | 40mg of MitoQ
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 1/15 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | 20mg of MitoQ (N=15) | 40mg of MitoQ (N=14)
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Had fall while taking recycling bin outside, the sun shone very bright in eyes and fell on side and injured nose. Did not seek medical attention and healed on own. Has been very light sensitive as a preexisting condition.
Cold (General disorders) | 1 | 0 | 0 — Cold Like symptoms
Hot Flashes (Reproductive system and breast disorders) | 0 | 1 | 0 — Had hot flashes after study started. Similar episode in the past while on estradiol patch.
Flu (General disorders) | 0 | 0 | 1 — Flu like symptoms

LIMITATIONS AND CAVEATS:
While the original sample size was 60 we were able to enroll only 45 subjects out of which 43 completed all visits. The study was affected due to COVID-19 and OHSU/VA contract delays.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04267926/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT04267926/ICF_000.pdf